CLINICAL TRIAL: NCT01219426
Title: A Transversal Study for the French Validation of Two Assessment Tools of Gambling Related Cognitions.
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Other Study IDs: 08/3-F
Record Dates: First submitted 2010-10-12; First posted 2010-10-13 (Estimated); Last update posted 2011-05-20 (Estimated); Status verified 2011-05

CONDITIONS: Gambling
Keywords: Gambling; cognitive distortions; assessment tool; validation; French
MeSH Terms: conditions — Gambling

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- students from the University of Nantes: To be more than 18 years old (the legal age to gamble in France)
  Interventions: Other: Filling of three questionnaires
- pathological gamblers seeking treatment: To be more than 18 years old (the legal age to gamble in France)and pathological gambler
  Interventions: Other: Filling of three questionnaires

INTERVENTIONS:
Other: Filling of three questionnaires — The only intervention of the study was the completion of the three questionnaires, and of a mini-questionnaire assessing gender, age, and gambling activities.

SUMMARY:
This study is divided into two stages. In the first stage, students from the University of Nantes completed the two assessment tools of gambling related cognitions (GABS : Gambling Attitudes and Beliefs Survey ; GRCS : Gambling Related Cognitions Scale), and a reference tool for gambling problem severity (SOGS : South Oaks Gambling Screen). In the second stage, consecutive pathological gamblers seeking treatment at the University Hospital of Nantes completed the three questionnaires. Only questionnaires from participants who reported gambling at least one time in the past year were kept for analyses.Responses of students gamblers and pathological gamblers presenting for treatment have been compiled for analysis.The main objective of the study is to validate the French adaptations of the GABS and the GRCS, and to explore their psychometric properties and structures.

DETAILED DESCRIPTION:
This study is divided into two stages. In the first stage, students from the University of Nantes completed the two assessment tools of gambling related cognitions (GABS : Gambling Attitudes and Beliefs Survey ; GRCS : Gambling Related Cognitions Scale), and a reference tool for gambling problem severity (SOGS : South Oaks Gambling Screen).

In the second stage, consecutive pathological gamblers seeking treatment at the University Hospital of Nantes completed the three questionnaires.

Only questionnaires from participants who reported gambling at least one time in the past year were kept for analyses.

Responses of students gamblers and pathological gamblers presenting for treatment have been compiled for analysis.

The main objective of the study is to validate the French adaptations of the GABS and the GRCS, and to explore their psychometric properties and structures.

The recruitment period for the first stage is comprised between March 2008 and August 2008.

The recruitment period for the second stage started in September 2008.

ELIGIBILITY:
Inclusion Criteria:

* To be more than 18 years old (the legal age to gamble in France)

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: To be more than 18 years old (the legal age to gamble in France)
Sampling Method: Non-Probability Sample
Dates: Start 2008-03; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marie Grall-Bronnec, MD, Principal Investigator — Nantes University Hospital
Locations (1):
- Nantes University Hospital, Nantes, France